CLINICAL TRIAL: NCT04580680
Title: Extracorporeal Blood Purification Therapy in Critically Ill Patients: an Interactive,Web-based,Multicenter,Observational Prospective Registry
Brief Title: Extracorporeal Blood Purification Therapy in Critically Ill Patients (GlobalARRT)
Acronym: GlobalARRT
Status: Recruiting | Type: Observational
Sponsor: Careggi Hospital (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Gianluca Villa, Principal investigator, Careggi Hospital
Other Study IDs: GlobalARRT
Record Dates: First submitted 2020-09-03; First posted 2020-10-08 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Critical Illness; Acute Kidney Injury; Sepsis; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Commercial membrane for Extracorporeal Blood Purification Therapy (EBPT) — At each participating center, EBP treatments with commercial membranes will be delivered in accordance with local practice and local levels of expertise. Enrolled patients will not receive additional treatments other than those routinely administered in ICUs. Nonetheless, all parameters settings for EBP treatments will be recorded in the web-based registry and analyzed a posteriori to reveal potential correlations with patient outcomes.

SUMMARY:
Worldwide, the use of Extracorporeal Blood Purification (EBP) in everyday clinical practice is becoming increasingly common, particularly in critical care settings. The efficacy of most of these treatments on removal of inflammatory mediators is the main rationale behind the use of EBP in critically ill patients with multiorgan dysfunction. Nonetheless, there are still some doubts as to the clinical efficacy of bacterial toxins and cytokines removal and many clinical trials aiming at exploring the effect of EBP on long-term outcomes of septic patients have failed to demonstrate consistent results regarding 28 day- or hospital-mortality rates. The primary aim of this observational prospective web-based registry is to define the possible clusters of critically ill patients - treated with extracorporeal blood purification therapies worldwide - who are homogeneous regarding both clinical and treatment characteristics and seem to benefit the most from EBP.

DETAILED DESCRIPTION:
Since May 2019, our research group has developed, implemented, and nationally spread the "ARRT registry" with the aim to describe the subpopulations of critically ill patients that benefit the most from EBP therapy with oXiris (6). The project is currently ongoing, involving more than 50 centers in Italy, with data from more than 65 patients treated with oXiris. Differently from other registries, the ARRT registry runs on a web-based platform easily accessible from internet-based technologies, including smartphones, that offers a user-friendly approach, facilitates data uploading, and enhances research collaboration. Furthermore, it adopts a proactive approach, in the sense that it includes several automatic calculators and decision support tools that might help clinicians to personalize treatments directly at the bedside (e.g. automatic calculation of clinical scoring systems, ideal body weight, mechanical ventilation setting, antibiotic adjustment according to renal function, etc.). All these tools can provide the clinician with real-time feedbacks. This web-based registry provides a clear example of translational medicine and translational research where data from clinical practice feed a database for clinical research and, contemporaneously, the database research tools improve clinical practice. Finally, this web-based registry allows each participating center to instantaneously evaluate its own data and obtain real-time basic statistics for each recorded variable (e.g. age at enrollment, main comorbidities, baseline serum creatinine, mortality rate, rate of multidrug-resistant bacteria, etc.), thus allowing for continuous monitoring of outcomes and local practices.

Overall, these features may prove particularly useful during treatment of critically ill septic patients with multiorgan dysfunction. Recently, the COVID-19 pandemic has been characterized by high prevalence of patients with severe multiorgan dysfunction, high mortality rate, lack of ICU resources, and the need for ICU discharge in a rapid, but safe, manner. The association between acute kidney injury and COVID-19 infection is well established. Organ crosstalk and systemic inflammation are the most accredited causes of Acute Kidney Injury (AKI) in these patients. Several EBP therapies have been proposed to attenuate systemic inflammation and/or support renal function in COVID-19 patients. Nevertheless, no data is currently available on application and feasibility of EBP therapies in COVID-19 patients or on their outcomes. Notably, the ARRT registry was able to effectively capture clinical data on systemic inflammation, organ dysfunction, and outcomes in patients treated with oXiris during the COVID-19 pandemic in Italy. In this regard, the implementation of a similar registry at the global level might prove effective for supporting clinicians involved in the treatment of patients with COVID-19 infection and multiorgan dysfunction worldwide.

ELIGIBILITY:
Inclusion Criteria: patients who meet all the following inclusion criteria may be included in this study:

1. Admission to ICU
2. Indications for at least one of the following extracorporeal blood purification treatments:

   1. Continuous Renal Replacement Therapy (CRRT) / Intermittent Hemodialysis (IHD) / Hybrid therapies for renal support/replacement;
   2. Immunomodulation therapy in critically ill patients using hemodiafilters with larger pore sizes characterized by enhanced transmembrane clearance of larger molecules (such as cytokines), hemodiafilters with enhanced unselective absorption of cytokines and/or endotoxins, cartridges with enhanced absorption of cytokines and/or endotoxins, techniques aimed at improving extracorporeal removal of cytokines and/or endotoxins.

It should be underlined that the lack of established guidelines on the use of membranes for extracorporeal blood purification (and on RRTs in general) leads to variability in clinical practice and treatments are initiated in accordance with the judgement of the responsible physician. Under these circumstances, it is preferable to keep inclusion criteria as wide as possible so as to obtain a real picture of clinical practice worldwide.

Exclusion Criteria: besides contraindications to the use of the EBP adopted (as from the manual of instructions), there are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All medical institutions that provide EBP treatments to critically ill patients are eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Define the possible clusters of critically ill patients | 10 days after Extracorporeal Blood Purification Therapy (EBPT) initiation
  Define the possible clusters of critically ill patients - treated with extracorporeal blood purification therapies worldwide - that are homogeneous regarding both clinical and treatment characteristics thanks all the treatment and baseline clinical variables extracted from the patient Case Report Forms (CRFs).

SECONDARY OUTCOMES:
To assess the correlation between cluster membership and positive short-term outcome. | 48 hours after EBPT initiation
  Define as ≥ 20% decrease in Vasoactive-Inotropic Score (VIS) at 48 hours with respect to baseline to assess the correlation between cluster membership and positive short-term outcome (i.e. an improvement in hemodynamic stability and inflammatory status).
To assess the correlation between cluster membership and positive long-term outcome. | 10 days after EBPT initiation
  To assess the correlation between cluster membership and positive long-term outcome, defined as patient survival at ICU discharge.
To assess the correlation between positive short-term outcome and changes from baseline. | 24 hours after EBPT initiation
  To assess the correlation between positive short-term outcome and changes from baseline in clinical parameters and all treatment at 12 and 24 hours (as from the patient CRFs).
To describe the clinical circumstances under which clinicians opt for specific techniques of extracorporeal blood purification therapy worldwide. | 10 days after EBPT initiation
  Timing of initiation of a specific Extracorporeal Blood Purification (EBT) treatment will be described.
To describe the clinical circumstances under which clinicians opt for specific techniques of extracorporeal blood purification therapy worldwide in terms of absolute and relative frequencies of clinical variables. | 10 days after EBPT initiation
  Absolute and relative frequencies of those clinical variables relevant to the application of a specific EBP treatment will be described.
To describe EBP utilization rates in intensive care units worldwide. | 10 days after EBPT initiation
  EBP utilization will be described in terms of cumulative incidence among all the enrolled patients from all participating centers
To describe EBP utilization rates in intensive care units worldwide in terms of absolute frequency | 10 days after EBPT initiation
  EBP utilization will be described in terms of of yearly absolute frequencies and cumulative incidence among all the enrolled patients from all participating centers.
To describe EBP in terms of relative frequencies for treatment type in intensive care units worldwide. | 10 days after EBPT initiation
  Utilization of Continuous Renal Replacement Therapy(CRRT), Intermittent Hemodialysis (IHD), and Hybrid Renal Replacement Therapies as well as of the different membranes will be described in terms of relative frequencies.
To describe EBP in terms of technical characteristics in intensive care units worldwide. | 10 days after EBPT initiation
  For each EBP treatment will be described absolute and relative frequency of chosen anticoagulation strategy
To describe EBP in terms of average flow rates in intensive care units worldwide. | 10 days after EBPT initiation
  For each EBP treatment will be described average flow rates (variables: blood flow rate, dialysate flow rate, replacement flow rate pre-filter, replacement flow rate post-filter, effluent flow rate, net ultrafiltration rate).

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Villa, md, Principal Investigator — University of Florence, Florence, Italy
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz DN, Antonelli M, Fumagalli R, Foltran F, Brienza N, Donati A, Malcangi V, Petrini F, Volta G, Bobbio Pallavicini FM, Rottoli F, Giunta F, Ronco C. Early use of polymyxin B hemoperfusion in abdominal septic shock: the EUPHAS randomized controlled trial. JAMA. 2009 Jun 17;301(23):2445-52. doi: 10.1001/jama.2009.856. PMID 19531784
- [Background] Klein DJ, Foster D, Schorr CA, Kazempour K, Walker PM, Dellinger RP. The EUPHRATES trial (Evaluating the Use of Polymyxin B Hemoperfusion in a Randomized controlled trial of Adults Treated for Endotoxemia and Septic shock): study protocol for a randomized controlled trial. Trials. 2014 Jun 11;15:218. doi: 10.1186/1745-6215-15-218. PMID 24916483
- [Background] Payen DM, Guilhot J, Launey Y, Lukaszewicz AC, Kaaki M, Veber B, Pottecher J, Joannes-Boyau O, Martin-Lefevre L, Jabaudon M, Mimoz O, Coudroy R, Ferrandiere M, Kipnis E, Vela C, Chevallier S, Mallat J, Robert R; ABDOMIX Group. Early use of polymyxin B hemoperfusion in patients with septic shock due to peritonitis: a multicenter randomized control trial. Intensive Care Med. 2015 Jun;41(6):975-84. doi: 10.1007/s00134-015-3751-z. Epub 2015 Apr 11. PMID 25862039
- [Background] Cutuli SL, Artigas A, Fumagalli R, Monti G, Ranieri VM, Ronco C, Antonelli M; EUPHAS 2 Collaborative Group. Polymyxin-B hemoperfusion in septic patients: analysis of a multicenter registry. Ann Intensive Care. 2016 Dec;6(1):77. doi: 10.1186/s13613-016-0178-9. Epub 2016 Aug 8. PMID 27502196
- [Background] Friesecke S, Trager K, Schittek GA, Molnar Z, Bach F, Kogelmann K, Bogdanski R, Weyland A, Nierhaus A, Nestler F, Olboeter D, Tomescu D, Jacob D, Haake H, Grigoryev E, Nitsch M, Baumann A, Quintel M, Schott M, Kielstein JT, Meier-Hellmann A, Born F, Schumacher U, Singer M, Kellum J, Brunkhorst FM. International registry on the use of the CytoSorb(R) adsorber in ICU patients : Study protocol and preliminary results. Med Klin Intensivmed Notfmed. 2019 Nov;114(8):699-707. doi: 10.1007/s00063-017-0342-5. Epub 2017 Sep 4. PMID 28871441
- [Background] Villa G, De Rosa S, Samoni S, Neri M, Cosimo C, Romagnoli S, Gavagni M, Ronco C, De Gaudio AR. oXirisNet Registry: A Prospective, National Registry on the oXiris Membrane. Blood Purif. 2019 Apr 11;47 Suppl 3:1-8. doi: 10.1159/000499356. Online ahead of print. PMID 30974438